CLINICAL TRIAL: NCT02426866
Title: The Risk of Cardiovascular Events Among HIV Patients Initiating Efavirenz-containing Versus Efavirenz-free Antiretroviral Regimens
Brief Title: Risk of CV Events With EFV vs. EFV-free Regimens
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Truven health (Unknown)
Responsible Party: Sponsor
Other Study IDs: AI266-414
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — efavirenz

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient with Efavirenz exposure: Patient with Efavirenz exposure
  Interventions: Drug: Efavirenz
- Patient without Efavirenz exposure: Patient without Efavirenz exposure
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz

SUMMARY:
The purpose of this study is to determine whether there is an increased risk of cardiovascular events (CV) with regimens containing efavirenz (EFV) versus other regimens in patients with HIV.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Aged 18 years or older on the index date
* Have at least one pharmacy claim for efavirenz or a drug in the comparison cohort during the period spanning January 1, 2007 through December 31,2013.
* Clinical Modification (ICD-9) diagnosis code for HIV infection including 042 (HIV disease), V08 (asymptomatic HIV infection status), 795.71 (nonspecific serologic evidence of HIV), and 079.53 (HIV, type 2) any time prior to the index claim.
* Have at least 6 months (180 days) of continuous enrollment prior to the index claim

Exclusion Criteria:

* Patients who have been dispensed any antiretroviral medications anytime before the index date including the 180-day baseline period
* Patients with evidence of a cardiovascular outcome of interest during the 180-day baseline period

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial insurance database and Medicaid database
Sampling Method: Non-Probability Sample
Enrollment: 29612 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events specifically based on incidence rate and compare the hazard between the HIV infected patient initiating efavirenz-containing antiretroviral regimen and efavirenz-free antiretroviral regimen | upto 1 to 5 years
  cardiovascular events specifically based on incidence rate and compare the hazard (myocardial infarction, stroke,percutaneous coronary intervention, coronary artery bypass graft, and composite of aforementioned events) between the HIV infected patient initiating efavirenz-containing antiretroviral regimen and efavirenz-free antiretroviral regimen

REFERENCES:
- See also: Related Info — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Related Info — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx